CLINICAL TRIAL: NCT00158860
Title: An International, Randomized, Double-Blind, Placebo-Controlled, Multicenter, 6-Month Study of the Efficacy and Safety of Valtrex 1g QD vs. Placebo for the Suppression of HSV-2 Genital Herpes in Newly Diagnosed Immunocompetent Patients
Brief Title: A Study Comparing Daily Treatment With Valaciclovir To Placebo For Suppression Of Herpes Simplex Virus HSV-2 Genital Herpes In Newly Diagnosed Patients. VALTREX® Tablet is a Trademark of the GlaxoSmithKline Group of Companies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS2100275
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2017-12

CONDITIONS: Herpes Genitalis
Keywords: VALTREX®; valaciclovir; genital herpes; HSV-2; suppression
MeSH Terms: conditions — Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valaciclovir (Experimental): Participants received double blinded treatment of oral dose of Valacyclovir 1 g given as 2 x 500 mg caplets QD for 6 months (24 weeks).
  Interventions: Drug: Valaciclovir
- Placebo (Placebo Comparator): Participants received double blinded treatment of oral dose of matching placebo to Valacyclovir 1 gram (g) given as 2 x 500 milligram (mg) caplets once daily (QD) for 6 months (24 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valaciclovir — 1g once daily
  Arms: Valaciclovir
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Genital herpes (GH) is a commonly occurring sexually transmitted disease caused by herpes simplex virus (HSV). There are two types of HSV, type 1 (HSV-1) and type 2 (HSV-2); both can cause GH, although the latter is much more likely to produce frequent recurrences of GH lesions. Evidence suggests that there are advantages to using suppressive vs. episodic treatment, which include increased intervals between the pain and discomfort of genital herpes recurrences. Therefore, this study will collect safety and efficacy data on suppressive therapy with valaciclovir in subjects newly diagnosed with HSV-2 genital herpes.

ELIGIBILITY:
Inclusion criteria:

* In overall general good health.
* Females can enter and participate in this study if they are of non-childbearing potential (i.e., physiologically incapable of becoming pregnant) or if of childbearing potential, has a negative pregnancy test (urine) at screening and agrees to use GSK stipulated contraceptive methods.
* Must be newly diagnosed with a first recognized episode of GH at the time of the Screening Visit or within 3 months prior to the Screening Visit.

Exclusion criteria:

* Known or suspected to be immunocompromised (e.g., subjects receiving immunosuppressive therapy or chemotherapy for malignancy, or are seropositive for HIV).
* Received an investigational drug in the 30 days prior to the study.
* Receiving systemic antiviral or immunomodulatory treatments.
* Must not have received systemic antiviral treatments (e.g., valaciclovir, Famvir (famciclovir), acyclovir, lysine) within 3 days of starting study drug or immunomodulatory treatments in the 30 days before starting study drug.
* Clinically significant impaired renal function as defined by a creatinine clearance <30 ml/min, calculated using the Cockcroft-Gault formula.
* Clinically significant impaired hepatic function defined as an ALT (alanine transaminase) level > 5 times the normal upper limit.
* Subjects with active liver disease.
* Known to be hypersensitive to acyclovir, famciclovir, ganciclovir or any component of valaciclovir formulations.
* Known resistance to acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir or valganciclovir.
* Subjects with malabsorption or vomiting syndrome or other gastrointestinal dysfunction that might impair drug pharmacokinetics.
* Women contemplating pregnancy within the duration of the study drug dosing period.
* Women who are pregnant and/or nursing mothers
* Current history of alcohol or drug abuse.
* Received suppressive (daily) therapy for genital herpes prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2004-06-21 (Actual); Primary Completion 2006-07-26 (Actual); Study Completion 2006-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (53):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Davis, California
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - GSK Investigational Site, Venice, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Alpharetta, Georgia
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Endicott, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Waukesha, Wisconsin
- GSK Investigational Site, Buenos Aires, Argentina
- Brazil (2):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Rio de Janeiro
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Québec
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HS2100275 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 74 centers in the Unites States, Canada, Argentina, Brazil, and Chile.
Pre-assignment Details: A total of 384 participants with first recognized episode of genital herpes (GH) were randomized in this study, out of which one participant did not take the study medication, hence, the Intent-to-treat (ITT) population consisted of 383 participants.
Groups:
- Placebo: Participants received double blinded treatment of oral dose of matching placebo to valacyclovir 1 gram (g) given as 2 x 500 milligram (mg) caplets once daily (QD) for 6 months (24 weeks). Participants with GH recurrences during the study temporarily discontinued their blinded treatment assignment and received open label valaciclovir 500 mg twice a day (BID) for 3 days after which the double-blind therapy was resumed.
- Valaciclovir 1g QD: Participants received double blinded treatment of oral dose of Valacyclovir 1 g given as 2 x 500 mg caplets QD for 6 months (24 weeks). Participants with GH recurrences during the study temporarily discontinued their blinded treatment assignment and received open label valaciclovir 500 mg BID for 3 days after which the double-blind therapy was resumed.
Period: Overall Study
Arm/Group | Placebo | Valaciclovir 1g QD
Started | 128 | 255
Completed | 93 | 184
Not Completed | 35 | 71
Not completed — Adverse Event | 3 | 6
Not completed — Lost to Follow-up | 11 | 17
Not completed — Protocol Violation | 8 | 23
Not completed — Withdrawal by Subject | 7 | 17
Not completed — MOVING OUT OF STATE | 1 | 0
Not completed — Pregnancy | 3 | 3
Not completed — SPONSOR STOPPED STUDY | 2 | 2
Not completed — SPONSOR REQUEST | 0 | 1
Not completed — Lost to Follow up but returned per GSK | 0 | 1
Not completed — Closed per sponsor | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants randomized to this treatment arm received matching placebo to valacyclovir 1 g given as 2 x 500 mg caplets QD for 6 months (24 weeks). Participants with GH recurrences during the study temporarily discontinued their blinded treatment assignment and received open label valaciclovir 500 mg BID for 3 days after which the double-blind therapy was resumed.
- Valaciclovir 1g QD: Participants received double blinded treatment of oral dose of valacyclovir 1 g given as 2 x 500 mg caplets QD for 6 months (24 weeks). Participants with GH recurrences during the study temporarily discontinued their blinded treatment assignment and received open label valaciclovir 500mg BID for 3 days after which the double-blind therapy was resumed.
- Total: Total of all reporting groups
Arm/Group | Placebo | Valaciclovir 1g QD | Total
Number analyzed (Participants) | 128 | 255 | 383
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (11.52) | 30.9 (10.48) | 31.3 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 176 | 268
  Male | 36 | 79 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Hispanic | 17 | 34 | 51
  Race: Arabic/North African | 0 | 2 | 2
  Race: Black | 39 | 84 | 123
  Race: East & South East Asian | 0 | 2 | 2
  Race: White/Caucasian | 68 | 125 | 193
  Race: Unknown | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Time to First GH Recurrence
Description: Diary cards were issued to the participants during randomization visit for recording GH recurrences. HSV recurrences since the last visit was assessed after review of the diary card and discussion with the participant. The percentage of participants with time to first GH recurrence was based on Kaplan-Meier estimates. Confidence intervals for differences in proportions was calculated using the standard error for the Kaplan-Meier estimate derived using Greenwood's formula.
Time Frame: Day 168
Population: ITT population was defined as all participants randomized to treatment who were administered at least one dose of investigational product.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo: Participants received double blinded treatment of oral dose of matching placebo to Valacyclovir 1 g given as 2 x 500 mg caplets QD for 6 months (24 weeks). Participants with GH recurrences during the study temporarily discontinued their blinded treatment assignment and received open label valaciclovir 500 mg BID for 3 days after which the double-blind therapy was resumed.
Arm/Group | Placebo | Valaciclovir 1g QD
Number analyzed (Participants) | 128 | 255
Percentage of participants | 43 | 71
Statistical Analysis 1: Comparison: Placebo vs Valaciclovir 1g QD; Test type: Superiority; p < 0.001, Log Rank; Kaplan-Meier estimates = 27.3, 95% CI 2-sided [16.0 to 38.6]
Statistical Analysis 2: Comparison: Placebo vs Valaciclovir 1g QD; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.401, 95% CI 2-sided [0.282 to 0.570]

2. Secondary Outcome: Mean Number of GH Recurrences Per Month Within the 6-month Study Period
Description: Mean number of GH recurrence reaching macular/papular stage per month was reported. Diary cards were issued to the participants during randomization visit for the recording GH recurrences. HSV recurrences since the last visit was assessed after review of the diary card and discussion with the participant.
Time Frame: Up to Day 168
Population: ITT population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Number of recurrences
Arm/Group | Placebo | Valaciclovir 1g QD
Number analyzed (Participants) | 122 | 227
Number of recurrences | 0.48 (1.860) | 0.11 (0.254)
Statistical Analysis 1: Comparison: Placebo vs Valaciclovir 1g QD; Test type: Superiority or Other; p < 0.001, Wilcoxon rank sum test

3. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE was defined as any untoward medical occurrence that, at any dose results in death, was life-threatening, required hospitalization or prolongation of hospitalization, results in disability/incapacity, was a congenital anomaly/birth defect or medically significant.
Time Frame: Upto Day 168
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Valaciclovir 1g QD
Number analyzed (Participants) | 128 | 255
Participants
  Any AEs | 98 | 185
  Any SAEs | 4 | 3

4. Secondary Outcome: Percentage of Participants With Time to First Oral Herpes Simplex Virus (HSV) Outbreak Within 6-months
Description: Diary cards were issued to the participants during randomization visit for recording HSV outbreak within 6-momths. HSV outbreak was assessed after review of the diary card and discussion with the participant. The percentage of participants who had first oral HSV outbreak at 6-months was reported.
Time Frame: Day 168
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Valaciclovir 1g QD
Number analyzed (Participants) | 128 | 255
Percentage of participants | 11 | 14

5. Secondary Outcome: Number of Isolates With Resistance to Acyclovir (ACV)
Description: Culture samples were tested for AVC-susceptibility by the analytical laboratory. Re-testing of the ACV resistant isolates was carried out to check if the half maximal inhibitory concentration (IC-50s) for all the ACV resistant isolates were within the expected errors of 2.0 microgram per milliliters (mcg/ml) cut-off for the plaque reduction assay. Those isolates that confirm to be resistant in repeat assays were considered as resistant to ACV.
Time Frame: Day 168
Population: ITT population.
Measure: Number; unit: Number of isolates
Arm/Group | Placebo | Valaciclovir 1g QD
Number analyzed (Participants) | 128 | 255
Number of isolates | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to end of study (Day 168).
Description: ITT population was defined as all participants randomized to treatment who were administered at least one dose of investigational product. ITT population was used for reporting adverse event.
Arm/Group | Placebo | Valaciclovir 1g QD
All-Cause Mortality (participants affected / at risk) | 0/128 | 1/255
Serious Adverse Events (participants affected / at risk) | 4/128 | 3/255
Other Adverse Events (participants affected / at risk) | 75/128 | 138/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | Valaciclovir 1g QD (N=255)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=128) | Valaciclovir 1g QD (N=255)
Nasopharyngitis (Infections and infestations) | 13 | 35
Herpes simplex (Infections and infestations) | 8 | 22
Vulvovaginal mycotic infection (Infections and infestations) | 12 | 16
Urinary tract infection (Infections and infestations) | 9 | 7
Influenza (Infections and infestations) | 7 | 7
Headache (Nervous system disorders) | 39 | 59
Dysmenorrhoea (Reproductive system and breast disorders) | 11 | 16
Nausea (Gastrointestinal disorders) | 10 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.